CLINICAL TRIAL: NCT01654133
Title: Evaluation of Visceral Function Following Endovascular Aortic Aneurysm Repair Using Branched Stent- Grafts
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: UNC Hospitals (Unknown); Cook Group Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 12-0644
Record Dates: First submitted 2012-07-27; First posted 2012-07-31 (Estimated); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Aortic Aneurysm, Abdominal; Ascending Aorta Aneurysm; Aortic Arch Aneurysm
Keywords: Aortic Aneurysm, abdominal; Ascending Aorta Aneurysm; Aortic Arch Aneurysm
MeSH Terms: conditions — Aortic Aneurysm, Abdominal; Aneurysm, Ascending Aorta; Aneurysm, Aortic Arch

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Endovascular TAAA Repair (Experimental): Endovascular repair of thoracoabdominal aortic aneurysm (TAAA) using Branched stent grafts
  Interventions: Device: Endovascular repair of thoracoabdominal aortic aneurysm (TAAA) using branched stent graft
- Endovascular Ascending/Aortic Arch Branch Repair (Experimental): Endovascular repair of aortic ascending/arch aneurysm using branched stent grafts
  Interventions: Device: Endovascular repair of ascending/arch aortic aneurysm using branched stent graft

INTERVENTIONS:
Device: Endovascular repair of thoracoabdominal aortic aneurysm (TAAA) using branched stent graft — Repair of thoracoabdominal aortic aneurysms
  Other Names: Endovascular repair of thoracoabdominal aortic aneurysm
  Arms: Endovascular TAAA Repair
Device: Endovascular repair of ascending/arch aortic aneurysm using branched stent graft — Repair of ascending/arch aortic aneurysms
  Other Names: Endovascular repair of ascending/ arch aortic aneurysm
  Arms: Endovascular Ascending/Aortic Arch Branch Repair

SUMMARY:
The purpose of this study is to evaluate visceral function, after endovascular repair of thoracoabdominal aneurysms or ascending/aortic arch aneurysms.

DETAILED DESCRIPTION:
This study will evaluate the effect of endovascular repair of thoracoabdominal aortic aneurysms (Types I-IV) on visceral function or aortic arch aneurysms using custom manufactured and off the shelf stent grafts. Specifically, the device orientation and configuration will be evaluated with respect to renal function. Since detailed CT scan imaging will be performed prior to and after endovascular repair, critical data concerning each branched vessel length, tangential orientation from the aorta, angle of incidence, and diameter can be determined. This information can then be coupled with hemodynamic data obtained from duplex ultrasonography as well as changes in renal volume, estimated glomerular filtration rate (eGFR), and flow characteristics over time. By analyzing the data in this fashion, it may be possible to determine changes in hemodynamics and/or physiologic conditions with respect to branched stent-graft design characteristics. These data may be utilized to enhance current device design and improve patient outcomes. The FDA has approved the use of commercially available devices to be used in conjunction with the investigational device if the Investigator deems this necessary.

ELIGIBILITY:
Cohort 1 (TAAA) Inclusion Criteria:

Patients may be included in the study if the patient has at least one of the following and has aortic anatomy appropriate for treatment with the Zenith® p-Branch™, Zenith® t-Branch, or Physician Specified TAAA Endovascular Graft (Custom Manufactured Devices).

1. Aortic Aneurysm Diameter

   a. TAAA (Type I - IV) (including pararenal subtypes) with orthogonal aortic diameter greater than or equal to 5 cm or b. greater than two times the normal aortic diameter
2. Rapid aortic enlargement (> than or equal to 5mm in 1 year)
3. Presence of a saccular aneurysm at risk for rupture based on investigators evaluation
4. Iliac artery aneurysm ˃2.2 cm may be treated with the Zenith® Branch Endovascular Graft-Iliac Bifurcation when the iliac artery aneurysm is associated with the qualifying thoracoabdominal aneurysm treated in this study

Exclusion Criteria:

General Exclusion Criteria

Patients must be excluded from the study if any of the following conditions are true:

1. Less than 18 years of age
2. Unwilling to comply with the follow-up schedule
3. Inability or refusal to give informed consent

Medical Exclusion Criteria

Patients must be excluded from the study if any of the following conditions are true:

1) Known sensitivities or allergies to stainless steel, nitinol, polyester, solder (tin, silver), polypropylene, urethane or gold 2) History of anaphylactic reaction to contrast material that cannot be adequately premedicated 3) Leaking, ruptured aneurysm associated with hypotension 4) Uncorrectable coagulopathy

Anatomical Exclusion Criteria

Patients must be excluded from the study if any of the following conditions are true:

1. Inadequate femoral/iliac access compatible with the required delivery systems;
2. Does not have a non-aneurysmal aortic segment proximal to the aneurysm with:

   a. A length of at least 4 mm, i.e. at least 4 mm circumferential wall contact around the limits of scallop b. A diameter measured outer wall to outer wall of no greater than 31mm and no less than 21 mm; c. An angle less than 60 degrees relative to the centerline of the aneurysm; d. An angle less than 45 degrees relative to the supraceliac aorta.
3. Does not have visceral vessel anatomy compatible with Zenith® p-Branch™, specifically:

   a. Renal vessel origins as measured relative to the superior mesenteric artery (SMA) compatible with the renal fenestration, i.e. Both renal vessel origins within 7.5mm of the corresponding renal fenestrations; b. Celiac vessel origin as measured relative to the superior mesenteric artery (SMA) compatible with the celiac scallop.
4. A proximal seal site with unsuitable thrombus/atheroma
5. Does not have iliac artery fixation sites and anatomy consistent with:

   1. Common iliac artery fixation site diameter, measured outer wall to outer wall on a sectional image (CT) <8.0 mm (prior to deployment)
   2. Iliac artery diameter, measured outer wall to outer wall on a sectional image (CT) >21 mm at distal fixation site
   3. Iliac artery distal fixation site <10 mm in length
   4. Inability to preserve at least one hypogastric artery

      -

Cohort 2 (ascending/aortic arch) Inclusion Criteria:

General Inclusion Criteria:

1. Treatment not possible with a currently available non-modified approved device
2. Patient accepts to and is able to comply with lifetime follow-up
3. Patient accepts to and is able to provide informed consent prior to enrollment
4. No stroke with significant residual deficit or myocardial infarction within the last 12 months
5. No significant carotid bifurcation disease (> 70% stenosis by NASCET criteria)
6. Absence of systemic or local infection that may increase the risk of endovascular graft infection
7. Patient determined to be a high-risk profile for open surgical repair considering any of the following items:

   1. Anatomy: previous sternotomy or left-sided thoracotomy (if the proposed open repair would require dissection of the thoracic aorta), previous aortic surgery, large aneurysm abutting the sternum with risk of disruption during sternotomy, prior cervical or chest irradiation.
   2. Physiology: ASA Category ≥ III, age >70 years, previous myocardial infarction, coronary artery disease, or coronary artery stent, coronary stress test with a reversible perfusion defect, COPD, congestive heart failure

Vascular Inclusion Criteria:

1. Aortic Aneurysm Diameter: Ascending and/or Arch aneurysm with or without aortic or aortoiliac aneurysm with orthogonal aortic diameter greater than two times the normal aortic diameter
2. Rapid aortic enlargement (≥ 5 mm in 1 year)
3. Presence of a saccular aneurysm at risk for rupture based on the investigators evaluation
4. Clinical indication for aneurysm repair based on symptoms
5. Concomitant thoracoabdominal and aortic arch aneurysm meeting one of the above-mentioned criteria.

Anatomic Inclusion Criteria:

1) There is enough space for the device to be deployed distal to coronary arteries and any coronary artery bypass grafts that are considered patent and necessary for proper cardiac perfusion 2) Ascending aortic length >50 mm (greater curve distance from sinotubular junction to proximal aspect of the innominate artery) 3) Sealing zone in the ascending aorta >40 mm in length and <38 mm in diameter for native aorta (<42 mm if surgical graft replacement in place) 4) Sealing zone in the great vessels of >20 mm in length

* Diameter of innominate artery used for sealing < 20 mm
* Diameter of CCA or subclavian artery used for sealing < 16mm 5. Distal aortic fixation zone: Native aorta or surgical graft (endovascular device or Dacron graft) , diameter: 20-42mm, distal neck length ≥20mm 6) Access for device delivery to accommodate 22F or 24F sheath depending on device design.

  7) Sealing zone in the great vessels of ≥ 20 mm in length
* Diameter of innominate artery used for sealing between 8 and 20 mm
* Diameter of CCA or subclavian artery used for sealing between 6 and 16 mm.

Extra inclusion criteria - special situations:

* Aortic dissection:

  1. A true lumen size large enough for device deployment and to gain access into the target branches
  2. A sealing zone in the target aorta (or surgical graft) that is proximal to the primary dissection, so that the graft would seal off the dissection lumen
  3. A sealing zone in the target supra-aortic trunk vessels that is distal to the dissection or surgically created
  4. Access into the true lumen from the groin and to at least one supra-aortic trunk vessel
* If more distal disease is observed in the aorta

  1. The repair might be coupled with a thoracoabdominal branched device
  2. Iliac anatomy large enough to allow the delivery of the arch branch device which is loaded within a 20F-24F sheath. Iliac conduits may be set in place if necessary.

Exclusion Criteria:

General exclusion criteria:

1. Life expectancy less than 2 years
2. Less than 18 years of age
3. Women must not be pregnant or breastfeeding
4. Active malignancy with life expectancy less than 2 years
5. Presence of mycotic aneurysm, systemic or local infection in access sites that may increase the risk of endovascular graft infection
6. Untreatable coagulopathy
7. Coronaropathy / Unstable angina
8. Anaphylactic reaction to contrast that cannot be adequately pre-medicated
9. Cultural objection to receipt of blood or blood products
10. Allergy or sensitivity to the endografts material (stainless steel, polyester, polypropylene, solder (tin, silver), gold, or nitinol)
11. Leaking or ruptured aneurysm associated with hypotension
12. Participation in another investigational clinical or device trial, except for participation in another investigational endovascular stent-graft protocol, percutaneous aortic valve protocol, or concomitant clinical trials designed to evaluate medical therapy strategies to reduce perioperative risk during fenestrated-branched endovascular repair
13. Prior open surgical or interventional procedure within 30 days of the anticipated date of the fenestrated-branched procedure, with the exception of planned procedures to provide access for repair (e.g. staged iliac conduit, cervical debranching) or to facilitate the procedure.

Anatomic Exclusion Criteria for the Cook Ascending/Arch graft

1. Significant occlusive disease, tortuosity, or calcification that would prevent endovascular access.
2. Iliac artery diameter, measured inner wall to inner wall on a sectional image (CT) <7.0 mm at any point along access length (prior to deployment). Inability to perform a temporary or permanent open surgical or endovascular iliac conduit for patients with inadequate femoral/iliac access.
3. Proximal seal length < 40 mm
4. Proximal seal site with a circumferential thrombus/atheroma/calcium

   -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 645 (Estimated)
Dates: Start 2012-07; Primary Completion 2035-08 (Estimated); Study Completion 2035-08 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in renal function over time (up to two years) after endovascular aortic aneurysm repair various custom stent grafts | Pre-procedure and 1, 6, 12, 18, and 24 months post procedure
  Visceral function after endovascular repair of pararenal aneurysms using various custom stent grafts. Specifically, the device orientation and configuration will be evaluated with respect to renal function over time. Critical data concerning each branched vessel from radiological studies coupled with hemodynamic data obtained from renal artery duplex, changes in renal volume, eGFR, and flow characteristics at 1, 6, 12, 18 and 24 months post procedure may make it possible to determine changes in renal function.

SECONDARY OUTCOMES:
Time to morbidity | 30 days and 1 & 2 years post procedure
  Morbidity at 30 days, 1 & 2 years post procedure
Time to mortality | 30 days and 1 & 2 years post procedure
  Mortality at 30 days, 1 & 2 years post procedure.
Time to loss of stent graft integrity | 30 days and 1 & 2 years post procedure
  Evidence on contrast CT angiography of loss of stent graft integrity at 30 days, and one and two years post procedure.
Time to migration | 30 days and 1 & 2 years post procedure
  Evidence of stent graft migration on abdominal x-rays at 30 days and 1 & 2 years.
Endoleak | 30 days and 1 & 2 years post procedure
  Evidence of Endoleak on contrast CT angiography of abdomen 30 days and 1 & 2 years post procedure.
Branch vessel Events | 30 days and 1 & 2 years post procedure
  Evidence of branch vessel events on contrast CT angiography and renal duplex 30 days, and 1 & 2 years post procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Mark A Farber, MD, Principal Investigator — University of North Carolina, Chapel Hill, NC 27599
Locations (1):
- UNC Heart and Vascular, Chapel Hill, North Carolina, United States

REFERENCES:
- [Derived] Mesnard T, Huang Y, Schanzer A, Timaran CH, Schneider DB, Mendes BC, Eagleton MJ, Farber MA, Parodi FE, Gasper WJ, Beck AW, Sweet MP, Zetterval SL, Lee A, Oderich GS; United States Aortic Research Consortium. Multicenter Prospective Evaluation of Patient Radiation Exposure During Fenestrated-Branched Endovascular Aortic Repair: A Ten-year Experience. Ann Surg. 2025 Feb 18. doi: 10.1097/SLA.0000000000006676. Online ahead of print. PMID 39963789
- [Derived] Oderich GS, Huang Y, Harmsen WS, Tenorio ER, Schanzer A, Timaran CH, Schneider DB, Mendes BC, Eagleton MJ, Farber MA, Gasper WJ, Beck AW, Sweet MP, Lee WA; United States Aortic Research Consortium. Early and Late Aortic-Related Mortality and Rupture After Fenestrated-Branched Endovascular Aortic Repair of Thoracoabdominal Aortic Aneurysms: A Prospective Multicenter Cohort Study. Circulation. 2024 Oct 22;150(17):1343-1353. doi: 10.1161/CIRCULATIONAHA.123.068234. Epub 2024 Jul 11. PMID 38989575
- [Derived] Finnesgard EJ, Beck AW, Eagleton MJ, Farber MA, Gasper WJ, Lee WA, Oderich GS, Schneider DB, Sweet MP, Timaran CH, Simons JP, Schanzer A; United States Aortic Research Consortium. Severity of acute kidney injury is associated with decreased survival after fenestrated and branched endovascular aortic aneurysm repair. J Vasc Surg. 2023 Oct;78(4):892-901. doi: 10.1016/j.jvs.2023.05.034. Epub 2023 Jun 16. PMID 37330702
- [Derived] Aucoin VJ, Motyl CM, Novak Z, Eagleton MJ, Farber MA, Gasper W, Oderich GS, Mendes B, Schanzer A, Tenorio E, Timaran CH, Schneider DB, Sweet MP, Zettervall SL, Beck AW; U.S. Aortic Research Consortium. Predictors and outcomes of spinal cord injury following complex branched/fenestrated endovascular aortic repair in the US Aortic Research Consortium. J Vasc Surg. 2023 Jun;77(6):1578-1587. doi: 10.1016/j.jvs.2023.01.205. Epub 2023 Apr 13. PMID 37059239